CLINICAL TRIAL: NCT05781295
Title: Multicentre Randomised Study Comparing a Taurolidine Lock and a Standard Saline Lock in the Primary Prevention of Catheter-related Endoluminal Infection in Paediatric Oncology.
Brief Title: Multicentre Randomised Study Comparing a Taurolidine Lock and a Standard Saline Lock in Paediatric Oncology
Acronym: PEDIALOCK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IC 2017-12
Record Dates: First submitted 2023-03-01; First posted 2023-03-23 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-07

CONDITIONS: Children; Medical Device; Primary Prevention; Oncology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TauroLock™ (Experimental): The patient will be followed up to a maximum of 6 months after randomization after have a Taurlock™ injected each time catheter will be used.
  Interventions: Device: TaurolockTM
- Physiological serum (NaCl 0.9%) (Placebo Comparator): The patient will be followed up to a maximum of 6 months after randomization after have a Physiological serum injected each time catheter will be used.
  Interventions: Device: Physiological serum

INTERVENTIONS:
Device: TaurolockTM — The patient will be followed up to a maximum of 6 months after randomization after have a TaurolockTM injected each time catheter will be used.
  Arms: TauroLock™
Device: Physiological serum — The patient will be followed up to a maximum of 6 months after randomization after have a Physiological serum injected each time catheter will be used.
  Arms: Physiological serum (NaCl 0.9%)

SUMMARY:
Interest of a Taurolidine lock at each catheter closure in the primary prevention of catheter-related endoluminal infection in paediatric oncology.

Multicentric, controlled, randomized and double-blind label study.

DETAILED DESCRIPTION:
The patient will be followed according to the type of pathology and the respective treatment protocol either Taurolock or physiological serum at each time cathter will be used.

ELIGIBILITY:
Inclusion Criteria:

1. Patient less than or equal to 21 years of age at inclusion.
2. Patient for whom a central catheter is planned to be inserted*, excluding a non-tunneled femoral or cervical external catheter or a peripherally inserted central catheter (as PICC line). *1st catheter placement or placement following a relapse (this placement must take place at least one month after previous catheter removal).
3. Patient treated for a cancer.
4. Patient with regular follow-up in the inclusion center.
5. Informed consent signed by the patient if adult or by legal representatives if minor.
6. Patient benefiting from a social security coverage.
7. Time between the date of catheter placement and the planned date for the first solution lock injection less than 6 weeks.

Exclusion Criteria:

1. Patient with retinoblastoma.
2. Allografted patient.
3. Patient with a life expectancy of less than 6 months.
4. Patient refusing to participate in the protocol.
5. Patient already receiving a central venous catheter-related infection prevention lock (ILCVC).
6. Patient with known allergy to citrate or (cyclo)-Taurolidine.
7. Patient taking other drugs with a known contraindication with citrate or (cyclo)-Taurolidine.
8. Patient with an external femoral catheter.
9. Patient with a PICCLINE-type peripheral venous inserted central catheter.
10. Patient unable to submit to the medical follow-up of the trial for geographical, social or psychological reasons.
11. Patient under guardianship and curatorship.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 148 (Estimated)
Dates: Start 2024-01-19 (Actual); Primary Completion 2028-07-23 (Estimated); Study Completion 2028-07-23 (Estimated)

PRIMARY OUTCOMES:
Comparison of the incidence of catheter-related infection per 1000 catheter days. | 1000 catheter days
  Comparison of the incidence of catheter-related infection per 1000 catheter days.

SECONDARY OUTCOMES:
Incidence of catheter colonizations. | through study completion, an average of 56 months
  Incidence of catheter colonizations.
Catheter removal time related to catheter complication. | through study completion, an average of 56 months
  Catheter removal time related to catheter complication.
Incidence of catheter removal related to catheter complication. | through study completion, an average of 56 months
  Incidence of catheter removal related to catheter complication.
Incidence of local infections (with or without bacteremia). | through study completion, an average of 56 months
  Incidence of local infections (with or without bacteremia).
Incidence of catheter occlusions. | through study completion, an average of 56 months
  Incidence of catheter occlusions.
Incidence of thrombotic complications. | through study completion, an average of 56 months
  Incidence of thrombotic complications.
Number and hospitalization duration related to catheter complications. | through study completion, an average of 56 months
  Number and hospitalization duration related to catheter complications.
Number and frequency of adverse events linked to lock. | through study completion, an average of 56 months
  Number and frequency of adverse events linked to lock.
Identification of microbiologic germs found in the hemocultures and catheter cultures after catheter removal for catheter infection. | through study completion, an average of 56 months
  Identification of microbiologic germs found in the hemocultures and catheter cultures after catheter removal for catheter infection.

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Institut Curie, Paris
  - Saint Louis, Paris
  - Armand Trousseau, Paris
  - Robert Debre, Paris
  - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: Yes
Sponsor will share de-identified data sets. Documents generated under the project will be disseminated in accordance with Institut Curie policies.
Supporting Information: Study Protocol, SAP
Time Frame: Data requests can be submitted starting 9 months after last article publication and will be made accessible for up to 12 months.
Access Criteria: Access to trial individual participant data can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a data sharing agreement (DSA).